CLINICAL TRIAL: NCT00738049
Title: A Phase 2, Investigator-Initiated, Feasibility Study to Evaluate the Mechanisms of Coronary Endothelial Dysfunction Imaged As Resting Myocardial Perfusion Heterogeneity After Endothelin Receptor Blockade With Darusentan
Brief Title: Darusentan Effect on PET Uptake Heterogeneity
Acronym: Darusentan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: K.Lance Gould (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, K.Lance Gould, Martin Bucksbaum distinguished University chair, Professor of Cardiovascualr MEdicine and Executive Director, Weatherhead P.E.T. Center for Preventing and Reversing Atherosclerosis, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-08-0380
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease; Endothelial Dysfunction
Keywords: atherosclerosis; coronary artery disease; myocardial perfusion defect; endothelial dysfunction; endothelin receptor blockade
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — darusentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will receive oral darusentan 100mg for 2 weeks during Phase 1 then placebo for 2 weeks during Phase 2.
  Interventions: Drug: darusentan 100 mg
- Group 2 (Active Comparator): Group 2 will receive placebo for 2 weeks during Phase 1 then oral darusentan 100 mg for two weeks during Phase 2
  Interventions: Drug: darusentan 100 mg

INTERVENTIONS:
Drug: darusentan 100 mg — All subjects will receive oral darusentan 100 mg for a total of 2 weeks and placebo for 2 weeks.
  Other Names: darusentan; CID 177236; LU-135252; HMR-4005; 171714-84-4

SUMMARY:
The primary objective of this study is to test the hypothesis that myocardial perfusion heterogeneity, quantified by Markovian Homogeneity analysis of cardiac PET perfusion images, will improve in a quantitative manner after treatment with selective ETA receptor antagonist darusentan 100 mg per day for 2 weeks compared to baseline and post-treatment PET scans in clinically stable subjects with coronary atherosclerosis and/or risk factors.

DETAILED DESCRIPTION:
This 6-week, Phase 2, randomized, double-blind, crossover, investigator-initiated, single-center study will determine the feasibility of detecting the effect of darusentan 100 mg once daily on the extent of myocardial perfusion heterogeneity in subjects with documented CAD, as measured by cardiac PET imaging. Prior to the initiation of any study procedures, an Informed Consent Form and HIPAA Authorization will be reviewed and signed by each subject. Screening assessments and evaluations may be conducted over a period of not more than 4 weeks.

Following a baseline PET scan (PET 1) subjects will be randomized to one of two treatment groups (Group 1 or Group 2), and receive blinded treatment for a total of 4 weeks. The 4-week treatment period will have two phases, Phase 1 and Phase 2. Group 1 will receive darusentan 100 mg for 2 weeks during Phase 1, then placebo for 2 weeks during Phase 2. Group 2 will receive placebo for 2 weeks during Phase 1, then darusentan 100 mg for 2 weeks during Phase 2. Following 4 weeks of treatment with blinded study drug, subjects in both treatment groups will be withdrawn from study drug for an additional 2 weeks. Maximum darusentan exposure in this study will be 2 weeks, and maximum placebo exposure in this study will be 2 weeks. Adjustments to the number or dosage of concomitant medications required for study entry will not be permitted at any time during the study.

A physical exam will be done at baseline and week 6 as well as blood chemistry and hematology samples taken. Vital signs and any adverse events will be monitored at each visit.

Efficacy will be assessed through cardiac PET imaging. In total, four PET scans will be administered: the first at the Randomization Visit (PET 1, Week 0); the second at the conclusion of Phase 1 (PET 2, Week 2); the third at the conclusion of Phase 2 (PET 3, Week 4) and the fourth at the conclusion of the Withdrawal period (PET 4, Week 6).

Subjects will be instructed to take their study drug with or without food once daily at approximately the same time in the morning throughout the course of the study. Subjects will also be instructed to take all concomitant medications consistently and at the same time each day throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be competent to provide written informed consent. Subjects must sign an IRB approved ICF and HIPAA Authorization prior to the initiation of any study procedures. All men must be informed of the potential risks of testicular tubular atrophy and infertility associated with taking study drug, and queried regarding their understanding of the potential risks as described in the ICF.
2. Subjects must be greater than 18 years of age.
3. Female subjects must be surgically sterile or documented as post-menopausal for at least 2 years.
4. Subjects must have documented coronary artery disease as evidenced by previous myocardial infarction, interventional procedure, significant stenosis by cardiac catheterization, or an abnormal perfusion study.
5. Subjects must have an abnormal PET scan.

Exclusion Criteria:

1. Subjects with acute heart failure
2. Subjects with sustained or symptomatic hypotension (SBP 90 mmHg)
3. Subjects with uncontrolled hypertension (SBP of 170 mmHg or DBP of 100 mmHg) at Screening
4. Subjects with unstable angina pectoris
5. Subjects with acute myocardial infarction, stroke, transient ischemic attack, or coronary angioplasty within the last 6 months
6. Subjects with primary valvular disease
7. Subjects with significant vascular aneurysm
8. Subjects with a documented history of renal failure
9. Subjects with liver disease (total bilirubin 3 mg/dL or serum ALT or AST >2X ULN)
10. Subjects with active malignancy
11. Subjects with a fatal non-cardiovascular disease that they are expected to succumb to within 1 year
12. Female subjects that are pregnant or lactating
13. Female subjects with the potential for child-bearing
14. Female subjects being treated with hormone therapies
15. Subjects with uncontrolled diabetes mellitus
16. Subjects with diabetes with gastro paresis or severe neuropathy
17. Subjects with a history of substance abuse within the last 2 years
18. Subjects who have participated in a clinical study involving another investigational drug or device within 1 month of the Screening Visit
19. Subjects with known hypersensitivity or allergy to L-arginine, aminophylline, adenosine, or dipyridamole
20. Subjects who have a planned surgical procedure during the course of the study
21. Subjects taking herbal food supplements (L-carnitine, L-arginine or Ginko biloba)
22. Subjects with known active or dormant type 2 herpes simplex virus infections
23. Subjects with a contraindication to treatment with an ERA. Contraindications may include, but are not limited to, evidence of elevated liver function tests (e.g., aminotransferases >2X ULN) or an event defined as a serious adverse event attributed to previous treatment with an ERA
24. Subjects who are judged by the investigator to be ineligible for this study for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Lance Gould, MD, Principal Investigator — University of Texas Medical School at Houston; Nils Johnson, MD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- Weatherhead PET Center for Preventing and Reversing Atherosclerosis, UT Medical School, Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Verma S, Anderson TJ. Fundamentals of endothelial function for the clinical cardiologist. Circulation. 2002 Feb 5;105(5):546-9. doi: 10.1161/hc0502.104540. No abstract available. PMID 11827916
- [Background] Clarkson P, Celermajer DS, Powe AJ, Donald AE, Henry RM, Deanfield JE. Endothelium-dependent dilatation is impaired in young healthy subjects with a family history of premature coronary disease. Circulation. 1997 Nov 18;96(10):3378-83. doi: 10.1161/01.cir.96.10.3378. PMID 9396430
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. Circulation. 2000 Apr 25;101(16):1899-906. doi: 10.1161/01.cir.101.16.1899. PMID 10779454
- [Background] Halcox JP, Schenke WH, Zalos G, Mincemoyer R, Prasad A, Waclawiw MA, Nour KR, Quyyumi AA. Prognostic value of coronary vascular endothelial dysfunction. Circulation. 2002 Aug 6;106(6):653-8. doi: 10.1161/01.cir.0000025404.78001.d8. PMID 12163423
- [Background] Bugiardini R, Manfrini O, Pizzi C, Fontana F, Morgagni G. Endothelial function predicts future development of coronary artery disease: a study of women with chest pain and normal coronary angiograms. Circulation. 2004 Jun 1;109(21):2518-23. doi: 10.1161/01.CIR.0000128208.22378.E3. Epub 2004 May 10. PMID 15136498
- [Background] Bottcher M, Madsen MM, Refsgaard J, Buus NH, Dorup I, Nielsen TT, Sorensen K. Peripheral flow response to transient arterial forearm occlusion does not reflect myocardial perfusion reserve. Circulation. 2001 Feb 27;103(8):1109-14. doi: 10.1161/01.cir.103.8.1109. PMID 11222474
- [Background] Nesto RW, Lamas GA, Barry J. Paradoxical elevation of threshold to angina pectoris by cold pressor test in men with significant coronary artery disease. Am J Cardiol. 1989 Mar 15;63(11):656-9. doi: 10.1016/0002-9149(89)90246-4. PMID 2923057
- [Background] Kjaer A, Meyer C, Nielsen FS, Parving HH, Hesse B. Dipyridamole, cold pressor test, and demonstration of endothelial dysfunction: a PET study of myocardial perfusion in diabetes. J Nucl Med. 2003 Jan;44(1):19-23. PMID 12515871
- [Background] el-Tamimi H, Mansour M, Wargovich TJ, Hill JA, Kerensky RA, Conti CR, Pepine CJ. Constrictor and dilator responses to intracoronary acetylcholine in adjacent segments of the same coronary artery in patients with coronary artery disease. Endothelial function revisited. Circulation. 1994 Jan;89(1):45-51. doi: 10.1161/01.cir.89.1.45. PMID 8281679
- [Background] Johnson NP, Gould KL. Physiology of endothelin in producing myocardial perfusion heterogeneity: a mechanistic study using darusentan and positron emission tomography. J Nucl Cardiol. 2013 Oct;20(5):835-44. doi: 10.1007/s12350-013-9756-5. Epub 2013 Jul 11. PMID 23842710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects who had undergone prior PET studies were contacted by mailings after a preliminary chart review. They received information about the study and were asked if they were interested in taking part in the study. If interested a screening visit was scheduled to determine if they met other inclusion/exclusion criteria.
Pre-assignment Details: After signing consent, study participants who met preliminary study criteria, were asked to come for the first PET scan. If rest homogeneity was too high by PET, the patient was excluded from randomization; otherwise the patient was randomized to receive placebo or study drug. 40 participants enrolled and 20 excluded by PET as explained above.
Groups:
- Darusentan Then Placebo,: Patients were randomized to oral Darusentan 100mg for 14 days and then underwent cardiac PET imaging. They then received placebo for 14 days and underwent PET imaging, followed by a washout period of 14 days and completed the final cardiac PET scan. Patients and physicians were blinded to medication assignment.
- Placebo, Then Darusentan 100mg: Patients were randomized to oral placebo for 14 days, then underwent PET imaging. Study patients then received Darusentan 100mg for 14 days. The patients underwent cardiac PET imaging followed by a 14 day washout period and final PET scan. Patients and physicians were blinded to medication assignment.
Period: 1st Intervention(14 Days)
Arm/Group | Darusentan Then Placebo, | Placebo, Then Darusentan 100mg
Started | 13 | 7
Completed | 13 | 7
Not Completed | 0 | 0
Period: 2nd Intervention(14 Days)
Arm/Group | Darusentan Then Placebo, | Placebo, Then Darusentan 100mg
Started | 13 | 7
Completed | 13 | 7
Not Completed | 0 | 0
Period: Washout
Arm/Group | Darusentan Then Placebo, | Placebo, Then Darusentan 100mg
Started | 13 | 7
Completed | 13 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 received oral Darusentan 100mg during Phase 1 then placebo during Phase 2.
- Group 2: Group 2 received placebo during Phase 1 then oral Darusentan 100 mg during Phase 2.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change During Darusentan Treatment in the Markovian Homogeneity Number, a Value That Quantitates Myocardial Perfusion Heterogeneity
Description: Markovian homogeneity analysis characterizes an image produced by a PET scan by examining the probability that a pixel with a given intensity will have a neighbor with a different intensity. The homogeneity index ranges from >0 to 1, where a value near 0 represents an image with a high probability that neighboring pixels have intensity values that differ greatly, and a value near 1 represents an image with a high probability that neighboring pixels have similar intensity values.
Time Frame: 0, 2, 4, and 6 weeks
Population: Statistical analysis is exploratory, therefore not easily planned. A paired t-test with 40 subjects will provide approximately 89% power to test the null hypothesis of no change in the homogeneity number versus a two-sided alternative at alpha= 5%,if the true mean change is 0.15,e.g.,a homogeneity index of 0.5 at baseline and 0.65 after darusentan.
Measure: Mean (Standard Deviation); unit: No units
Groups:
- Baseline: All patients underwent a baseline assessment of Markovian homogeneity before receiving darusentan or placebo
- Darusentan 100mg: All patients underwent a baseline assessment of Markovian homogeneity while taking darusentan
Arm/Group | Baseline | Darusentan 100mg
Number analyzed (Participants) | 20 | 20
No units | 0.33 (0.04) | 0.39 (0.10)

2. Secondary Outcome: Change During Darusentan Treatment in Absolute Flow at Rest and Hyperemia
Time Frame: 0, 2, 4, and 6 weeks
Measure: Mean (Standard Deviation); unit: cc/min/gm
Groups:
- Darusentan 100mg at Rest: All patients underwent assessment of rest flow while receiving darusentan
- Darusentan 100mg at Hyperemia: All patients underwent assessment of hyperemic flow while receiving darusentan
- Baseline at Rest: All patients underwent a baseline assessment of resting flow before receiving darusentan or placebo
- Baseline at Hyperemia: All patients underwent a baseline assessment of hyperemic flow before receiving darusentan or placebo
Arm/Group | Darusentan 100mg at Rest | Darusentan 100mg at Hyperemia | Baseline at Rest | Baseline at Hyperemia
Number analyzed (Participants) | 20 | 20 | 20 | 20
cc/min/gm | 0.65 (0.13) | 1.97 (0.54) | 0.50 (0.10) | 2.03 (0.56)

3. Secondary Outcome: Change During Darusentan Treatment in the Coronary Flow Reserve (CFR)
Description: CFR is calculated as the unitless ratio between hyperemic to resting flow
Time Frame: 0, 2, 4, and 6 weeks
Measure: Mean (Standard Deviation); unit: no units
Groups:
- Baseline: All patients underwent a baseline assessment of CFR before receiving darusentan or placebo
- Darusentan 100mg: All patients underwent a assessment of CFR while receiving darusentan
Arm/Group | Baseline | Darusentan 100mg
Number analyzed (Participants) | 20 | 20
no units | 3.52 (0.80) | 3.04 (0.61)

ADVERSE EVENTS:
Groups:
- Group 1: Darusentan 100mg during Phase 1, Placebo during Phase 2
- Group 2: Received placebo during Phase 1, Darusentan 100mg during Phase 2
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7

LIMITATIONS AND CAVEATS:
The trial was stopped after 20 enrollments as the manufacturer of darusentan halted further development of the drug after a negative phase 3 trial in resistant hypertension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No